CLINICAL TRIAL: NCT03472430
Title: Randomized Controlled Trial of Transcutaneous Electrical Nerve Stimulation for Pain Relief During Transvaginal Oocyte Retrieval Using Conscious Sedation
Brief Title: Transcutaneous Electrical Nerve Stimulation During Transvaginal Oocyte Retrieval
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TENS TUGOR ver 1
Record Dates: First submitted 2018-02-25; First posted 2018-03-21 (Actual); Last update posted 2019-02-28 (Actual); Status verified 2019-02

CONDITIONS: Transcutaneous Electric Nerve Stimulation; Oocyte Retrieval
Keywords: Oocyte Retrieval; Transcutaneous Electric Nerve Stimulation; Pain relief; Conscious sedation
MeSH Terms: interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment group (Active Comparator): Transcutaneous electrical nerve stimulation machine, start 5 minutes before start of oocyte retrieval and stop 5 minutes after removal of oocyte retrieval needle
  Interventions: Device: Transcutaneous electrical nerve stimulation
- Placebo group (Sham Comparator): TENS machine with electrodes not emitting any impulses, start 5 minutes before start of oocyte retrieval and stop 5 minutes after removal of oocyte retrieval needle
  Interventions: Device: TENS machine with electrodes not emitting any impulses.

INTERVENTIONS:
Device: Transcutaneous electrical nerve stimulation — The TENS machine used in the study will be the Endomed 482 that delivers biphasic pulsed currents using pulse duration of 400 µs and pulse frequencies between 80-100 pulses.
  Other Names: Endomed 482
  Arms: Treatment group
Device: TENS machine with electrodes not emitting any impulses. — TENS machine with electrodes not emitting any impulses.
  Arms: Placebo group

SUMMARY:
This randomized double-blinded control trial aims to compare the pain levels experienced by the women using the standard conscious sedation and those who had transcutaneous electrical nerve stimulation (TENS) in addition to conscious sedation. The hypothesis is that there will be less pain in women with both conscious sedation and TENS.

DETAILED DESCRIPTION:
Women who are indicated to undergo IVF in our center will be assessed for eligibility for the study. Written consent will be obtained from those who agreed to join the study.

Eligible women recruited will be randomized according to a computer-generated randomization list prepared by a designated research staff into one of the two groups on the day of oocyte retrieval

1. Patient with both conscious sedation and active TENS
2. Patient with conscious sedation and placebo TENS

Blinding Both the women and the physician performing the procedure will be blinded from the group allocation.

Checking of effectiveness of blinding will be done by asking the patient and the physician after the procedure as to which group they think the women is in.

The procedure Women will receive ovarian stimulation according to the departmental Standard Operating Procedures. Ovarian stimulation will be monitored by ultrasound. Human chorionic gonadotrophin or an agonist (decapeptyl) will be given when the dominant follicle is at least 18mm and there are three more follicles of at least 16mm. Oocyte retrieval will then be arranged 36 hours later.

Prior to oocyte retrieval, two sets of self-adhesive electrodes will be placed on the women back on each side of the spine at T10 to S4 level. Instructions on how to titrate the TENS amplitude to the desired level that gives a strong non-painful electrical paraesthesia will be given to the women by the research nurse who is unaware of the group allocation. TENS therapy will start 5 minutes before the procedure and stop 5 minutes after the removal of oocyte aspiration needle. The TENS machine used in the study will be the Endomed 482 that delivers biphasic pulsed currents using pulse duration of 400 µs and pulse frequencies between 80-100 pulses s-. The women in the treatment group will be given a TENS machine with electrodes emitting impulses while those in the placebo group will be given a TENS machine with electrodes that is not emitting any impulses.

The woman lies on the operative bed in a lithotomy position. 25mg Pethidine and 5mg Diazepam will be given intravenously. The blood pressure and pulse of the woman are checked after the drug administration and the oxygen saturation is monitored continuously throughout the procedure. 10ml 1% lignocaine is injected to the paracervical region by the operating surgeon with a 21-gauge needle after cleansing the vagina and cervix with chlorhexidine. Under transvaginal ultrasound guidance, a 16-gauge ovum aspiration needle is introduced. Aspiration of follicles is performed with a suction pressure of 100 mmHg.

ELIGIBILITY:
Inclusion Criteria:

* Women who undergo transvaginal oocyte retrieval

Exclusion Criteria:

* There is only one ovary
* Oocyte retrieval performed on one ovary only
* There are less than three follicles >=16mm in diameter
* Allergic to pethidine or midazolam
* Previous experience with TENS
* Skin damage or allergy at site of TENS pads application
* History of pacemaker insertion

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 160 (Actual)
Dates: Start 2018-05-04 (Actual); Primary Completion 2018-10-15 (Actual); Study Completion 2018-10-15 (Actual)

PRIMARY OUTCOMES:
Pain level | 1 day on the day of the retrieval procedure
  The women will be asked to rate the pain according to a 100mm linear visual analogue scale. The visual analogue scale range from 0 to 100, 0 indicating no pain and 100 indicating maximum pain. A small value in the visual analogue scale indicates lower pain levels, therefore better. It is a single level indicated by the patients.

SECONDARY OUTCOMES:
Side effects | 1 day on the day of the retrieval procedure
  Side effects experienced by the women
Women satisfaction | 1 day on the day of the retrieval procedure
  Patient's satisfaction towards pain relief will be assessed before discharge. They will be rated as 5, 'excellent'; 4, 'satisfactory'; 3, 'fair'; 2,'not very satisfactory' and 1, 'totally unsatisfactory.

CONTACTS AND LOCATIONS:
Overall Officials: Ernest HY Ng, MD, Principal Investigator — The University of Hong Kong
Locations (1):
- Department of Obstetrics and Gynaecology, Hong Kong, Hong Kong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ng EH, Tang OS, Chui DK, Ho PC. A prospective, randomized, double-blind and placebo-controlled study to assess the efficacy of paracervical block in the pain relief during egg collection in IVF. Hum Reprod. 1999 Nov;14(11):2783-7. doi: 10.1093/humrep/14.11.2783. PMID 10548622
- [Background] Ng EH, Tang OS, Chui DK, Ho PC. Comparison of two different doses of lignocaine used in paracervical block during oocyte collection in an IVF programme. Hum Reprod. 2000 Oct;15(10):2148-51. doi: 10.1093/humrep/15.10.2148. PMID 11006189
- [Background] Ng EH, Chui DK, Tang OS, Ho PC. Paracervical block with and without conscious sedation: a comparison of the pain levels during egg collection and the postoperative side effects. Fertil Steril. 2001 Apr;75(4):711-7. doi: 10.1016/s0015-0282(01)01693-4. PMID 11287024
- [Background] Lier MC, Douwenga WM, Yilmaz F, Schats R, Hompes PG, Boer C, Mijatovic V. Patient-Controlled Remifentanil Analgesia as Alternative for Pethidine with Midazolam During Oocyte Retrieval in IVF/ICSI Procedures: A Randomized Controlled Trial. Pain Pract. 2015 Jun;15(5):487-95. doi: 10.1111/papr.12189. Epub 2014 Apr 12. PMID 24725465
- [Background] Kwan I, Bhattacharya S, Knox F, McNeil A. Pain relief for women undergoing oocyte retrieval for assisted reproduction. Cochrane Database Syst Rev. 2013 Jan 31;(1):CD004829. doi: 10.1002/14651858.CD004829.pub3. PMID 23440796
- [Background] Johnson M. Watson T. Transcutaneous electrical nerve stimulation, Electrotherapy: Evidence-based Practice. , 2008 Edinburgh Churchill Livingstone (pg. 253 -96)
- [Background] Santana LS, Gallo RB, Ferreira CH, Duarte G, Quintana SM, Marcolin AC. Transcutaneous electrical nerve stimulation (TENS) reduces pain and postpones the need for pharmacological analgesia during labour: a randomised trial. J Physiother. 2016 Jan;62(1):29-34. doi: 10.1016/j.jphys.2015.11.002. Epub 2015 Dec 11. PMID 26701166
- [Background] Lison JF, Amer-Cuenca JJ, Piquer-Marti S, Benavent-Caballer V, Bivia-Roig G, Marin-Buck A. Transcutaneous Nerve Stimulation for Pain Relief During Office Hysteroscopy: A Randomized Controlled Trial. Obstet Gynecol. 2017 Feb;129(2):363-370. doi: 10.1097/AOG.0000000000001842. PMID 28079781
- [Derived] Wong QHY, Lui MW, Yung SSF, Ko JKY, Li RHW, Ng EHY. Randomized controlled trial of transcutaneous electrical nerve stimulation for pain relief during transvaginal oocyte retrieval using conscious sedation: study protocol for a randomized controlled trial. Trials. 2019 Apr 11;20(1):205. doi: 10.1186/s13063-019-3227-5. PMID 30971304

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-11-24): https://cdn.clinicaltrials.gov/large-docs/30/NCT03472430/Prot_SAP_000.pdf